CLINICAL TRIAL: NCT00054925
Title: Weight Loss Maintenance (WLM)
Acronym: WLM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Pro00013066; U01HL068734 (NIH)
Record Dates: First submitted 2003-02-13; First posted 2003-02-14 (Estimated); Last update posted 2012-03-07 (Estimated); Status verified 2012-03

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Obesity; Diabetes Mellitus, Non-insulin Dependent; Hypertension
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Obesity; Diabetes Mellitus, Type 2; Hypertension

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Personal contact (PC) (Active Comparator): The Personal Contact (PC) intervention offers one-on-one guidance and support in maintaining weight loss.
  Interventions: Behavioral: Personal contact (PC)
- Interactive technology (IT) (Active Comparator): Utilizes internet and automated phone technology to enhance the frequency and timeliness of feedback.
  Interventions: Behavioral: Interactive technology (IT)

INTERVENTIONS:
Behavioral: Personal contact (PC) — This arm uses brief, individual contacts on a monthly basis which emphasize core elements of weight maintenance. Monthly contacts with an interventionist occur for 30 months after the end of Phase I. Face-to-face contacts occur approximately every four months (e.g., three annually), with telephone contacts occurring every month between FTF contacts.
  Arms: Personal contact (PC)
Behavioral: Interactive technology (IT) — The website utilizes collaborative goal setting and problem-solving strategies to identify contingent action plans for perceived obstacles to success. In order to tailor the intervention to the needs of the participant, the action plan can be updated anytime and as frequently as desired by the individual. Participants are encouraged to input data on weight, food records, physical activity, and goals on a weekly basis. Participants are not restricted to logging on to the website only once a week. Rather, participants have the option of logging on to the website to enter data, communicate with other participants, or to seek other information, as frequently as they wish.
  Arms: Interactive technology (IT)

SUMMARY:
To determine the effectiveness of continuous patient contact on weight loss maintenance.

DETAILED DESCRIPTION:
BACKGROUND:

Overweight/obesity is the second leading cause of death in the US, and is growing in prevalence at an alarming rate. Control of overweight/obesity is increasingly recognized as a high national priority because of its contribution to cardiovascular (CVD) risk factors and ultimately to CVD itself. The short-term success of behavioral interventions for weight loss has been repeatedly documented. Unfortunately, because weight re-gain is extremely common, a disappointingly, small proportion of individuals achieve long-term weight control. Of the factors that are associated with sustained weight loss, one of the most important is continued intervention with frequent contacts.

DESIGN NARRATIVE:

The study is a multi-center, randomized, controlled trial [Weight Loss Maintenance Trial (MAINTENANCE)] to determine the effects of two innovative behavioral interventions, each designed to maintain frequent contacts, compared to a usual care control group. Overweight and obese individuals (60% women, 40% African Americans) who are taking medication for hypertension, dyslipidemia and/or type 2 diabetes will enter a 6-month, weight loss program. Those 800 individuals who lose at least 4 kg (approximately 9 pounds) will then be randomized into one of three groups: a Personal Contact (PC) Intervention that provides monthly personal contacts with a trained interventionist, primarily via telephone; an Interactive Technology (IT) Intervention that provides frequent contacts through a state-of-the-art interactive web-based program supplemented by other communication technologies; or Usual Care (UC). The primary outcome will be weight change from the end of the initial weight loss program to the end of the 30-month weight maintenance intervention period. Other outcomes will include weight change in subgroups, prevalence of CVD risk factors, measures of behavior change, and cost of implementation. For each outcome, the Personal Contact and Interactive Technology interventions will be compared to Usual Care and, if different from Usual Care, to each other. To successfully combat the obesity epidemic, clinicians and health care systems must have options that are effective and feasible and that can be provided to large numbers of individuals.

Phase II intervention completed: July 2007

Phase III intervention completed: October 2009

ELIGIBILITY:
Overweight men and women who took medication for hypertension, type 2 diabetes and/or hyperlipidemia in the six month weight loss phase. and who were able to lose approximately 9 pounds. There will be approximately 60% women and 40% African Americans.

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1685 (Actual)
Dates: Start 2003-01; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Change in Weight | Baseline to 30 months

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Appel, Principal Investigator — Johns Hopkins University; Phillip Brantley, Principal Investigator — LSU Pennington Biomedical Research Center; Jack Hollis, Principal Investigator — Kaiser Foundation Research Institute; Victor Stevens, Principal Investigator — Kaiser Foundation Research Institute; Laura Svetkey, Study Chair — Duke University

REFERENCES:
- [Derived] Coughlin JW, Brantley PJ, Champagne CM, Vollmer WM, Stevens VJ, Funk K, Dalcin AT, Jerome GJ, Myers VH, Tyson C, Batch BC, Charleston J, Loria CM, Bauck A, Hollis JF, Svetkey LP, Appel LJ; Weight Loss Maintenance Collaborative Research Group. The impact of continued intervention on weight: Five-year results from the weight loss maintenance trial. Obesity (Silver Spring). 2016 May;24(5):1046-53. doi: 10.1002/oby.21454. Epub 2016 Mar 15. PMID 26991814
- [Derived] Coughlin JW, Gullion CM, Brantley PJ, Stevens VJ, Bauck A, Champagne CM, Dalcin AT, Funk KL, Hollis JF, Jerome GJ, Lien LF, Loria CM, Myers VH, Appel LJ. Behavioral mediators of treatment effects in the weight loss maintenance trial. Ann Behav Med. 2013 Dec;46(3):369-81. doi: 10.1007/s12160-013-9517-3. PMID 23813320
- [Derived] Batch BC, Shah SH, Newgard CB, Turer CB, Haynes C, Bain JR, Muehlbauer M, Patel MJ, Stevens RD, Appel LJ, Newby LK, Svetkey LP. Branched chain amino acids are novel biomarkers for discrimination of metabolic wellness. Metabolism. 2013 Jul;62(7):961-9. doi: 10.1016/j.metabol.2013.01.007. Epub 2013 Feb 1. PMID 23375209
- [Derived] Stolzenberg-Solomon RZ, Falk RT, Stanczyk F, Hoover RN, Appel LJ, Ard JD, Batch BC, Coughlin J, Han X, Lien LF, Pinkston CM, Svetkey LP, Katki HA. Sex hormone changes during weight loss and maintenance in overweight and obese postmenopausal African-American and non-African-American women. Breast Cancer Res. 2012 Oct 31;14(5):R141. doi: 10.1186/bcr3346. PMID 23113944
- [Derived] Myers VH, McVay MA, Champagne CM, Hollis JF, Coughlin JW, Funk KL, Gullion CM, Jerome GJ, Loria CM, Samuel-Hodge CD, Stevens VJ, Svetkey LP, Brantley PJ. Weight loss history as a predictor of weight loss: results from Phase I of the weight loss maintenance trial. J Behav Med. 2013 Dec;36(6):574-82. doi: 10.1007/s10865-012-9450-0. Epub 2012 Aug 21. PMID 22907176
- [Derived] Champagne CM, Broyles ST, Moran LD, Cash KC, Levy EJ, Lin PH, Batch BC, Lien LF, Funk KL, Dalcin A, Loria C, Myers VH. Dietary intakes associated with successful weight loss and maintenance during the Weight Loss Maintenance trial. J Am Diet Assoc. 2011 Dec;111(12):1826-35. doi: 10.1016/j.jada.2011.09.014. PMID 22117658
- [Derived] Funk KL, Stevens VJ, Appel LJ, Bauck A, Brantley PJ, Champagne CM, Coughlin J, Dalcin AT, Harvey-Berino J, Hollis JF, Jerome GJ, Kennedy BM, Lien LF, Myers VH, Samuel-Hodge C, Svetkey LP, Vollmer WM. Associations of internet website use with weight change in a long-term weight loss maintenance program. J Med Internet Res. 2010 Jul 27;12(3):e29. doi: 10.2196/jmir.1504. PMID 20663751
- [Derived] Svetkey LP, Stevens VJ, Brantley PJ, Appel LJ, Hollis JF, Loria CM, Vollmer WM, Gullion CM, Funk K, Smith P, Samuel-Hodge C, Myers V, Lien LF, Laferriere D, Kennedy B, Jerome GJ, Heinith F, Harsha DW, Evans P, Erlinger TP, Dalcin AT, Coughlin J, Charleston J, Champagne CM, Bauck A, Ard JD, Aicher K; Weight Loss Maintenance Collaborative Research Group. Comparison of strategies for sustaining weight loss: the weight loss maintenance randomized controlled trial. JAMA. 2008 Mar 12;299(10):1139-48. doi: 10.1001/jama.299.10.1139. PMID 18334689
- [Derived] Stevens VJ, Funk KL, Brantley PJ, Erlinger TP, Myers VH, Champagne CM, Bauck A, Samuel-Hodge CD, Hollis JF. Design and implementation of an interactive website to support long-term maintenance of weight loss. J Med Internet Res. 2008 Jan 25;10(1):e1. doi: 10.2196/jmir.931. PMID 18244892